CLINICAL TRIAL: NCT04858425
Title: A 2-Part, 2-Arm, Phase 2, Randomized, Double-Blind, Placebo-Controlled Study on the Safety and Efficacy of Niclosamide in Patients With COVID-19 With Gastrointestinal Infection
Brief Title: Safety and Efficacy of Niclosamide in Patients With COVID-19 With Gastrointestinal Infection
Acronym: RESERVOIR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The termination of the study was a decision based on topline data analysis (no efficacy as per Day 43) of the study data.
Sponsor: Entero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZ-NICL-COV-1
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2023-06

CONDITIONS: Covid19
Keywords: SARS-CoV-2; Covid; Covid19 Diarrhea; Covid19 GI Infection
MeSH Terms: conditions — COVID-19 | interventions — Niclosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Niclosamide (Experimental): Niclosamide tablets 400 mg 3 times daily for 14 days
  Interventions: Drug: Niclosamide
- Placebo (Placebo Comparator): Matching placebo tablets 3 times daily for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Niclosamide — Niclosamide tablets 400 mg 3 times daily for 14 days
  Arms: Niclosamide
Drug: Placebo — Matched placebo tablets 400 mg 3 times daily for 14 days
  Arms: Placebo

SUMMARY:
This is a 2-part, 2-arm, Phase 2 , multicentre, randomized, double-blind, placebo-controlled study in adults with COVID-19 with gastrointestinal infection.

ELIGIBILITY:
Inclusion Criteria:

1. Part 1 only, patients with a primary diagnosis of COVID-19, with or without pneumonia, who agree to be monitored daily for at least 7 days after randomization and who accept continuing to be assessed for the study procedures.
2. Part 2 only, patients with a primary diagnosis of COVID-19, with or without pneumonia.

Exclusion Criteria:

1. At the time of randomization, patients who require intensive care unit (ICU) admission or patients with severe respiratory insufficiency who require mechanical ventilation or with rapid worsening of respiratory function leading to expectation for mechanical ventilation or ICU admission.
2. Evidence of rapid clinical deterioration or existence of any life-threatening co-morbidity or any other medical condition that, in the opinion of the investigator, makes the patient unsuitable for inclusion.
3. Patients who, at the time of enrollment, are not in a clinical condition compatible with the oral administration of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2023-09-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (13):
  - Central Alabama Research, Birmingham, Alabama
  - Midland Florida Clinical Research Center, LLC, DeLand, Florida
  - New Generation Medical Research, Hialeah, Florida
  - LCC Medical Reserach Institute, LLC, Miami, Florida
  - Westchester General Hospital, Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - P & S Research, LLC, Miami, Florida
  - University of South Florida, Tampa, Florida
  - IACT Health - Roswell, Columbus, Georgia
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - Homestead Associates in Research, Homestead Meadows, Texas
  - SMS Clinical Research LLC, Mesquite, Texas
  - Tranquil Research, Webster, Texas
- India (7):
  - Yashoda Hospital, Secunderabad, Andhra Pradesh
  - SSG Hospital and Medical Institute, Vadodara, Gujarat
  - GMERS Medical College and Hospital, Vadodara, Gujarat
  - Noble Hospital Private Limited, Pune, Maharashtra
  - Sir Ganga Ram Hospital, Nagar, New Delhi
  - Maharaja Agrasen Superspeciality Hospital, Jaipur, Jaipur, Rajasthan
  - Malla Reddy Narayana Multispecialty Hospital, Hyderabad, Telangana
- Ukraine (5):
  - Communal Non-Commercial Medical Enterprise "Likarnya Prydniprovska", Kremenchuk, Poltava Oblast
  - Municipal Non-profit Enterprise "City Clinical Hospital # 4" of Dnipro City Council, Dnipro
  - Municipal Non-profit Enterprise Central City Clinical Hospital of Ivano-Frankivsk City Council, Ivano-Frankivsk
  - Municipal Non-Profit Enterprise City Clinical Hospital 13 of Kharkiv Regional Council, Kharkiv
  - Private Enterprise Private Manufacturing Company Acinus, Kropyvnytskyi

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Niclosamide | Placebo
Started | 84 | 82
Completed | 74 | 77
Not Completed | 10 | 5
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 4 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Niclosamide | Placebo | Total
Number analyzed (Participants) | 84 | 82 | 166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 77 | 74 | 151
  >=65 years | 7 | 8 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 46 | 93
  Male | 37 | 36 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 63 | 118
  Not Hispanic or Latino | 29 | 19 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 4 | 3 | 7
  Black or African American | 0 | 0 | 0
  White | 71 | 74 | 145
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: SAEs
Description: Serious adverse event (SAE) coded by System Organ Class (SOC) and Preferred Term (PT), using the Medical Dictionary for Regulatory Activities (MedDRA).
Time Frame: Day 1 to 6 weeks
Measure: Number; unit: participants
Arm/Group | Niclosamide | Placebo
Number analyzed (Participants) | 84 | 82
participants
  Infections and infestations | 0 | 1
  Injury, poisoning and procedural complications | 0 | 1

2. Primary Outcome: TEAE
Description: Proportion of patients with Treatment Emergent Adverse Events (TEAE) leading to study drug discontinuation.
Time Frame: Day 1 to 6 weeks
Measure: Number; unit: participants
Arm/Group | Niclosamide | Placebo
Number analyzed (Participants) | 84 | 82
participants
  Gastrointetinal disorders | 1 | 1
  Blood and lymphatic system disorders | 0 | 1
  Endocrine disorders | 0 | 1
  Infections and infestations | 0 | 1
  Injury, poisoning and procedural complications | 0 | 1
  Investigations | 1 | 1
  Musculoskeletal and connective tissue disorders | 0 | 1

3. Primary Outcome: Fecal RNA Virus Clearance
Description: Time to fecal viral RNA clearance (stool sample) assessed by RT-qPCR in the niclosamide arm compared to the placebo arm.
Time Frame: Day 1 to 6 weeks
Measure: Number; unit: participants
Arm/Group | Niclosamide | Placebo
Number analyzed (Participants) | 60 | 58
participants
  Day 4 | 8 | 9
  Day 8 | 21 | 20
  Day 15 | 40 | 33
  Day 22 | 48 | 42
  Day 29 | 51 | 43
  Day 36 | 51 | 45
  Day 43 | 52 | 48

4. Primary Outcome: Safety Laboratory Tests Including CBC, BUN, Blood Sugar, Electrolytes (Specifically Leukocytes and Platelets)
Description: Change in safety laboratory tests, including CBC, BUN, blood sugar, electrolytes, alkaline phosphatase, AST, ALT, LDH, total bilirubin, serum creatinine, from baseline to 6 weeks, the number of subjects with values low, normal, and high compared to the normal ranges pretreatment versus post-treatment will be provided.
Time Frame: Day 1 to Day 43
Measure: Median (Full Range); unit: cells (10^9/L)
Arm/Group | Niclosamide | Placebo
Number analyzed (Participants) | 78 | 79
cells (10^9/L)
  Leukocytes | 0.340 [-12.71 to 4.38] | 0.495 [-11.13 to 5.70]
  Platelets | 11.5 [-196 to 116] | 3.0 [-337 to 148]

5. Primary Outcome: Safety Laboratory Tests Including CBC, BUN, Blood Sugar, Electrolytes (Specifically Erythrocytes)
Description: Change in safety laboratory tests, including CBC, BUN, blood sugar, electrolytes, alkaline phosphatase, AST, ALT, LDH, total bilirubin, serum creatinine, from baseline to 6 weeks, the number of subjects with values low, normal, and high compared to the normal ranges pretreatment versus post-treatment will be provided.
  Erythrocytes
Time Frame: Day 1 to Day 43
Measure: Median (Full Range); unit: cells 10^12/L
Arm/Group | Niclosamide | Placebo
Number analyzed (Participants) | 78 | 79
cells 10^12/L | -0.250 [-0.87 to .85] | -0.125 [-0.96 to 0.84]

6. Primary Outcome: Safety Laboratory Tests Including CBC, BUN, Blood Sugar, Electrolytes (Specifically Hemocrit)
Description: Change in safety laboratory tests, including CBC, BUN, blood sugar, electrolytes, alkaline phosphatase, AST, ALT, LDH, total bilirubin, serum creatinine, from baseline to 6 weeks, the number of subjects with values low, normal, and high compared to the normal ranges pretreatment versus post-treatment will be provided.
  Hemocrit (L/L)
Time Frame: Day 1 to Day 43
Measure: Median (Full Range); unit: L/L
Arm/Group | Niclosamide | Placebo
Number analyzed (Participants) | 78 | 79
L/L | -0.0195 [-0.100 to 0.077] | -0.0130 [-0.141 to 0.072]

7. Primary Outcome: Safety Laboratory Tests Including CBC, BUN, Blood Sugar, Electrolytes (Specifically Hemoglobin)
Description: Change in safety laboratory tests, including CBC, BUN, blood sugar, electrolytes, alkaline phosphatase, AST, ALT, LDH, total bilirubin, serum creatinine, from baseline to 6 weeks, the number of subjects with values low, normal, and high compared to the normal ranges pretreatment versus post-treatment will be provided.
  Hemoglobin (g/L)
Time Frame: Day 1 to Day 43
Measure: Median (Full Range); unit: g/L
Arm/Group | Niclosamide | Placebo
Number analyzed (Participants) | 78 | 79
g/L | -4.0 [-30 to 13] | -2.5 [-39 to 14]

8. Primary Outcome: Safety Laboratory Tests Including CBC, BUN, Blood Sugar, Electrolytes (Specifically Corpuscular Volume)
Description: Change in safety laboratory tests, including CBC, BUN, blood sugar, electrolytes, alkaline phosphatase, AST, ALT, LDH, total bilirubin, serum creatinine, from baseline to 6 weeks, the number of subjects with values low, normal, and high compared to the normal ranges pretreatment versus post-treatment will be provided.
  Corpuscular volume (fL)
Time Frame: Day 1 to Day 43
Measure: Median (Full Range); unit: fL
Arm/Group | Niclosamide | Placebo
Number analyzed (Participants) | 78 | 79
fL | -0.35 [-10.5 to 9.3] | -0.75 [-16.1 to 15.8]

9. Primary Outcome: Safety Laboratory Tests Including CBC, BUN, Blood Sugar, Electrolytes (Specifically BUN, Glucose, Chloride, Potassium, and Sodium)
Description: as for outcome 4
Time Frame: Day 1 to Day 43
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Niclosamide | Placebo
Number analyzed (Participants) | 78 | 79
mmol/L
  BUN | 0.000 [-6.07 to 4.65] | 0.000 [-8.21 to 3.21]
  Glucose | -0.360 [-5.22 to 3.28] | 0.110 [-9.15 to 3.28]
  Chloride | 2.0 [-7 to 9] | 1.0 [-9 to 13]
  Potassium | 0.00 [-1.0 to 1.1] | 0.10 [-1.9 to 2.1]
  Sodium | 1.0 [-6 to 7] | 0.0 [-13 to 7]

10. Primary Outcome: Safety Laboratory Tests Including CBC, BUN, Blood Sugar, Electrolytes (Specifically Alkaline Phosphatase, AST, ALT, and LDH)
Description: as for outcome 4
Time Frame: Day 1 to Day 43
Measure: Median (Full Range); unit: U/L
Arm/Group | Niclosamide | Placebo
Number analyzed (Participants) | 78 | 79
U/L
  Alkaline Phosphatase | 2.0 [-173 to 26] | 2.0 [-76 to 49]
  AST | -2.5 [-117 to 98] | -1.0 [-151 to 26]
  ALT | -3.0 [-70 to 73] | -4.0 [-77 to 32]
  LDH | -2.0 [-209 to 157] | 6.0 [-86 to 102]

11. Primary Outcome: Safety Laboratory Tests Including CBC, BUN, Blood Sugar, Electrolytes (Specifically Bilirubin and Serum Creatinine)
Description: as for outcome 4
Time Frame: Day 1 to Day 43
Measure: Median (Full Range); unit: mcmol/L
Arm/Group | Niclosamide | Placebo
Number analyzed (Participants) | 78 | 79
mcmol/L
  Bilirubin | 0.60 [-10.7 to 10.1] | 1.20 [-4.3 to 22]
  Creatinine | 0.0 [-53 to 44] | 0.0 [-44 to 27]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Niclosamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/84 | 2/82
Other Adverse Events (participants affected / at risk) | 1/84 | 1/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niclosamide (N=84) | Placebo (N=82)
Infections and infestations (Infections and infestations) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niclosamide (N=84) | Placebo (N=82)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 1 (1)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Endocrine disorders (Endocrine disorders) | 0 (0) | 1 (1)
Infections and infestations (Infections and infestations) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Investigations (Investigations) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT04858425/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT04858425/SAP_001.pdf